CLINICAL TRIAL: NCT01884597
Title: Investigator Sponsored Trial of Polypoidal Choroidal Vasculopathy (PCV) Evaluation Assessing High-Dose Ranibizumab Prospectively
Brief Title: Investigator Sponsored Trial of Polypoidal Choroidal Vasculopathy (PCV) Evaluation Assessing High-Dose Ranibizumab Prospectively (PEARL2)
Acronym: PEARL2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hawaii Pacific Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Gregg T. Kokame, MD, Medical Director, The Retina Center at Pali Momi, Hawaii Pacific Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4929S
Record Dates: First submitted 2012-06-01; First posted 2013-06-24 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: PCV; Polypoidal Choroidal Vasculopathy
Keywords: PEARL2; PCV; Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Active Comparator): 12 monthly, intravitreal injections of 2.0mg ranibizumab followed by 12 monthly, intravitreal injections of 1.0mg ranibizumab
  Interventions: Drug: high-dose ranibizumab; Drug: ranibizumab
- Cohort 2 (Active Comparator): 6-months of monthly, intravitreal injections of ranibizumab 2.0mg followed by 18 months of monthly, intravitreal injections of ranibizumab 1.0mg
  Interventions: Drug: high-dose ranibizumab; Drug: ranibizumab
- Cohort 3 (Active Comparator): 24 months of monthly, intravitreal injections of ranibizumab 1.0mg
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: high-dose ranibizumab — 20mg ranibizumab vials, 0.05ml injected intravitreally, monthly
  Arms: Cohort 1; Cohort 2
Drug: ranibizumab — 3 mg ranibizumab, liquid, vials, 0.1ml injected intravitreally monthly
  Other Names: Lucentis

SUMMARY:
This is a 24-month study of ranibizumab (2.0 mg and 1.0 mg) in subjects with polypoidal choroidal vasculopathy as diagnosed by fluorescein/indocyanine green (FA/ICG) angiography.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 25 years
* Polypoidal choroidal vasculopathy as noted on fluorescein and ICG angiography: active leakage, active bleeding or recent decrease in vision
* BCVA using ETDRS of 20/32 to 20/400

Exclusion Criteria:

* Any history of previous vitrectomy
* Any prior treatment with verteporfin photodynamic therapy in the study eye.
* Previous cataract surgery within the preceding 2 months of Day 0
* Active intraocular inflammation in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease)
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
* Prior anti-vascular endothelial growth factor (VEGF) (Macugen, Avastin, Lucentis) in the study eye prior within 30 days prior to enrollment in this study
* Known allergy to any component of the study drug
* Blood pressure >180/110 (systolic above 180 or diastolic above 110) If blood pressure if brought below 180/110 by anti-hypertensive treatment, the patient can become eligible.
* Major surgery within 28 days prior to randomization or major surgery planned within the next 12 months. Major surgery is defined as a surgical procedure that is more extensive than needle biopsy/aspiration placement of a central venous access device, removal/biopsy of a skin lesion, or placement of a peripheral venous catheter.
* Myocardial infraction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 6 months prior to randomization.
* Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomization.
* History of recurrent significant infections or bacterial infections
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception, surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicide gel, an intra uterine device (IUD), or contraceptive hormone implant or patch
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial.

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg T Kokame, MD, MMM, Principal Investigator — Hawaii Pacific Health
Locations (3):
- United States (3):
  - Retina Consultants of Hawaii, Honolulu, Hawaii
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - The Retina Center at Pali Momi, ‘Aiea, Hawaii

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 24 months of monthly, intravitreal injections of ranibizumab 1.0mg
  ranibizumab: 1 mg/0.1 ml ranibizumab, liquid, vials, 0.1ml injected intravitreally monthly
- Cohort 2: 6-months of monthly, intravitreal injections of ranibizumab 2.0mg followed by 18 months of monthly, intravitreal injections of ranibizumab 1.0mg
  high-dose ranibizumab: 2.0mg/0.05ml ranibizumab, 0.05ml injected intravitreally, monthly
  ranibizumab: 1 mg/0.1 ml ranibizumab, liquid, vials, 0.1ml injected intravitreally monthly
- Cohort 3: 12 monthly, intravitreal injections of 2.0mg ranibizumab followed by 12 monthly, intravitreal injections of 1.0mg ranibizumab
  high-dose ranibizumab: 2.0mg/0.05ml ranibizumab, 0.05ml injected intravitreally, monthly
  ranibizumab: 1 mg/0.1 ml ranibizumab, liquid, vials, 0.1ml injected intravitreally monthly
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 5 | 3 | 16
Completed | 4 | 2 | 15
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 4 | 2 | 15 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 3 | 1 | 13 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.75 (13.72) | 71.00 (19.80) | 77.47 (8.37) | 77.17 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 5 | 7
  Male | 2 | 2 | 10 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 15 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 15 | 21

OUTCOME MEASURES:

1. Primary Outcome: BCVA
Description: Mean change in best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) eye chart at a starting test distance of 4 meters from Baseline to Month 12.
Time Frame: From Baseline to Month 12
Measure: Mean (Standard Deviation); unit: number of letters read correctly
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
number of letters read correctly | -3.50 (21.52) | 29.50 (24.75) | 8.60 (12.57)

2. Primary Outcome: BCVA
Description: Mean change in best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters from Baseline to Month 24
Time Frame: Baseline to M24
Measure: Mean (Standard Deviation); unit: number of letters read correctly
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
number of letters read correctly | -5.75 (24.58) | 23.5 (44.54) | 5.13 (15.98)

3. Secondary Outcome: Ocular Adverse Events (AE)
Description: Incidence and severity of ocular adverse events, as identified by eye examination (including visual acuity testing)
Time Frame: Monthly
Measure: Number; unit: Ocular adverse events
Groups:
- Cohort 1; Cohort 2; Cohort 3: No ocular adverse events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
Ocular adverse events | 0 | 0 | 0

4. Secondary Outcome: Systemic AEs
Description: Incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs
Time Frame: Monthly
Measure: Number; unit: Number of Participants with Systemic AEs
Groups:
- Cohort 1: 24 months of monthly, intravitreal injections of ranibizumab 1.0mg
  ranibizumab: 3 mg ranibizumab, liquid, vials, 0.1ml injected intravitreally monthly
- Cohort 3: 12 monthly, intravitreal injections of 2.0mg ranibizumab followed by 12 monthly, intravitreal injections of 1.0mg ranibizumab
  high-dose ranibizumab: 20mg ranibizumab vials, 0.05ml injected intravitreally, monthly
  ranibizumab: 3 mg ranibizumab, liquid, vials, 0.1ml injected intravitreally monthly
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
Number of Participants with Systemic AEs | 0 | 0 | 1

5. Secondary Outcome: BCVA
Description: Best corrected visual acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters, at Baseline, Day 14, Month 1, Month 3, Month 6, Month 9 , Month 12, Month 15, Month 18, Month 21 and Month 24
Time Frame: at Baseline, Day 14, Month 1, Month 3, Month 6, Month 9 , Month 12, Month 15, Month 18, Month 21 and Month 24
Measure: Mean (Standard Deviation); unit: number of letters read correctly
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
number of letters read correctly
  Baseline | 55.00 (19.06) | 50.00 (28.28) | 62.80 (17.11)
  Day 14 | 52.00 (18.92) | 52.50 (24.75) | 64.07 (18.47)
  Month 1 | 47.00 (27.83) | 70.00 (8.49) | 65.67 (16.60)
  Month 3 | 48.50 (32.60) | 78.50 (6.36) | 69.13 (18.19)
  Month 6 | 47.50 (31.65) | 82.50 (4.95) | 69.33 (15.43)
  Month 9 | 51.75 (32.90) | 72.50 (2.12) | 71.67 (9.64)
  Month 12 | 51.50 (33.16) | 79.50 (3.54) | 71.40 (10.66)
  Month 15 | 48.00 (34.97) | 80.50 (0.71) | 70.80 (10.35)
  Month 18 | 48.00 (32.38) | 83.00 (4.24) | 69.93 (10.91)
  Month 21 | 50.00 (33.34) | 67.50 (9.19) | 68.533 (12.14)
  Month 24 | 49.25 (31.92) | 73.50 (16.26) | 67.93 (13.08)

6. Secondary Outcome: Macular Edema
Description: Optical Coherence Tomography (OCT) central macular and peripapillary thickness
Time Frame: Baseline, Day 14, Month 1-24
Population: Patient in Cohort 2 missed several visits.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
microns
  Baseline | 370.25 (148.14) | 347.50 (194.45) | 282.47 (44.55)
  Day 14 | 265.00 (69.58) | 251.00 (65.05) | 235.07 (35.45)
  Month 1 | 276.25 (22.56) | 228.00 (24.04) | 216.67 (33.47)
  Month 2 | 252.50 (15.46) | 218.50 (14.85) | 212.20 (33.06)
  Month 3 | 244.25 (12.18) | 220.00 (12.73) | 216.29 (33.50)
  Month 4 | 238.25 (16.60) | 224.00 (15.56) | 214.36 (26.33)
  Month 5 | 245.75 (20.95) | 224.50 (12.02) | 215.53 (40.77)
  Month 6 | 232.75 (24.70) | 224.00 (9.90) | 211.47 (36.32)
  Month 7 | 234.00 (19.29) | 223.00 (12.73) | 215.67 (30.90)
  Month 8: number analyzed (Participants) | 4 | 1 | 15
  Month 8 | 233.00 (16.79) | 232.00 (NA) — One patient missed a visit. | 209.67 (34.01)
  Month 9 | 229.75 (17.93) | 222.50 (9.19) | 203.29 (31.04)
  Month 10: number analyzed (Participants) | 4 | 1 | 15
  Month 10 | 217.00 (7.00) | 233.00 (NA) — One patient missed a visit | 215.80 (30.05)
  Month 11 | 223.25 (19.87) | 228.50 (12.02) | 206.93 (32.04)
  Month 12 | 225.00 (18.22) | 226.50 (9.19) | 207.80 (29.33)
  Month 13 | 221.67 (17.16) | 222.00 (15.56) | 209.71 (39.34)
  Month 14 | 244.50 (34.32) | 223.00 (15.56) | 211.27 (32.19)
  Month 15 | 220.25 (17.56) | 228.50 (12.02) | 210.20 (29.27)
  Month 16 | 220.25 (20.71) | 227.5 (10.61) | 212.00 (31.18)
  Month 17: number analyzed (Participants) | 4 | 1 | 15
  Month 17 | 219.75 (22.51) | 238 (NA) — One patient missed a visit | 209.29 (31.94)
  Month 18 | 237075 (57.72) | 230.50 (14.85) | 213.67 (32.73)
  Month 19 | 218.33 (24.54) | 231.5 (9.19) | 217.08 (41.69)
  Month 20: number analyzed (Participants) | 4 | 1 | 15
  Month 20 | 216.00 (25.97) | 237 (NA) — Patient missed a visit | 217.93 (36.11)
  Month 21 | 214 (23.83) | 218.5 (17.68) | 209.07 (32.46)
  Month 22 | 211.5 (27.01) | 239.50 (12.02) | 212.13 (36.50)
  Month 23 | 209.25 (28.92) | 244.50 (21.92) | 216.08 (33.64)
  Month 24 | 214.25 (22.65) | 231.00 (1.41) | 215.27 (38.83)

7. Secondary Outcome: PCV Anatomic Changes
Description: Decrease and/or resolution in the branching vascular network of the PCV complex as measured by mean size of the branched vascular network (BVN) on ICG and fluorescein angiography
  Decrease and/or resolution of the polyps of the PCV complex as measured on ICG and fluorescein angiography
Time Frame: Baseline, Months 6, 12, 24
Measure: Number; unit: Participants with PCV Anatomic Changes
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 15 | 2 | 4
Participants with PCV Anatomic Changes
  Baseline (BVN) | 0 | 0 | 0
  Month 6 (BVN) | 0 | 0 | 1
  Month 12 (BVN) | 2 | 0 | 1
  Month 24 (BVN) | 1 | 0 | 2
  Baseline (PCV) | 0 | 0 | 0
  Month 6 (PCV) | 3 | 2 | 8
  Month 12 (PCV) | 2 | 1 | 8
  Month 24 (PCV) | 4 | 2 | 9

8. Secondary Outcome: Fundus Clinical Findings
Description: Decrease in subretinal hemorrhage or exudates as measured by mean size as noted on fundus photography and clinic exam
Time Frame: Baseline, Months 6, 12, 24
Measure: Number; unit: Participants with Fundus Findings
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 2 | 15
Participants with Fundus Findings
  Baseline | 0 | 0 | 0
  Month 6 | 1 | 2 | 8
  Month 12 | 1 | 2 | 8
  Month 24 | 1 | 2 | 8

ADVERSE EVENTS:
Time Frame: Adverse event data include events starting on day 0 and ending at month 24.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/2 | 0/15
Other Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=2) | Cohort 3 (N=15)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pneumonia requiring hospitalization. Adverse event recorded by follow up call and visits.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=3) | Cohort 3 (N=15)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) — Patient explained during visit.
Rash (General disorders) | 0 (0) | 0 (0) | 1 (2) — Patient explained during visit.
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Patient explained during visit.
Body ache, fever, hives (General disorders) | 0 (0) | 0 (0) | 1 (1) — Patient explained during visit
Bone Marrow Tap (Investigations) | 0 (0) | 0 (0) | 1 (1) — Patient explained during visit.
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Patient explained during visit.
Stent Placement for artery blockage (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Patient explained during visit.
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Patient explained during visit.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Patient explained during visit.

LIMITATIONS AND CAVEATS:
Small sample size for each arms group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No